CLINICAL TRIAL: NCT04377620
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Assess the Efficacy and Safety of Ruxolitinib in Participants With COVID-19-Associated ARDS Who Require Mechanical Ventilation (RUXCOVID-DEVENT)
Brief Title: Assessment of Efficacy and Safety of Ruxolitinib in Participants With COVID-19-Associated ARDS Who Require Mechanical Ventilation (RUXCOVID-DEVENT)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated by sponsor
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 18424-369
Expanded Access: NCT04355793 (No longer available)
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: Cytokine storm; COVID-19; ARDS; SARS-CoV-2; ruxolitinib; pneumonia
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome; Pneumonia | interventions — ruxolitinib; Janus Kinase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo + Standard of Care (SoC) (Placebo Comparator): Matching Placebo will be administered BID approximately 12 hours apart without regard to food/feeding via enteric feeding tube or oral.
  Interventions: Drug: Placebo
- Ruxolitinib 5mg + Standard of Care (SoC) (Experimental): Ruxolitinib 5mg will be administered BID approximately 12 hours apart without regard to food/feeding via enteric feeding tube or oral.
  Interventions: Drug: Ruxolitinib
- Ruxolitininb 15mg + Standard of Care (SoC) (Experimental): Ruxolitinib 15mg will be administered BID approximately 12 hours apart without regard to food/feeding via enteric feeding tube or oral.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Placebo — Placebo administered BID approximately 12 hours apart
  Arms: Placebo + Standard of Care (SoC)
Drug: Ruxolitinib — Ruxolitinb administered BID approximately 12 hours apart
  Other Names: INCB018424; Oral Jak Inhibitor
  Arms: Ruxolitinib 5mg + Standard of Care (SoC); Ruxolitininb 15mg + Standard of Care (SoC)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ruxolitinib in the treatment of participants with COVID-19-associated Acute Respiratory Distress Syndrome (ARDS) who require mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Participant or guardian health proxy must provide informed consent before any study assessment is performed.
* Male or female participants aged ≥ 12 years.
* Participants with coronavirus (SARS-CoV-2) infection confirmed ≤ 3 weeks prior to randomization by any test with local regulatory approval.
* Participants who are intubated and receiving mechanical ventilation due to COVID-19-associated ARDS and have a PaO2/FiO2 of ≤ 300 mmHg within 6 -hours of randomization.

Participants with lung imaging showing bilateral or diffuse pulmonary infiltrates on chest x-ray or CT scan.

Exclusion Criteria:

* Known history of hypersensitivity to any drugs or metabolites of similar chemical classes as ruxolitinib.
* Presence of severely impaired renal function defined by estimated creatinine clearance < 15 mL/min measured or calculated by Cockcroft-Gault equation or calculated by the updated bedside Schwartz equation. Participants must not be receiving CRRT or intermittent hemodialysis at screening.
* In the opinion of the investigator, unlikely to survive for > 24 hours from randomization.
* Suspected active uncontrolled bacterial, fungal, viral, or other infection (besides COVID-19).
* Currently receiving ECMO.
* Participant may not be sharing a ventilator, or co-ventilating, with any other patient.
* Treatment with anti-IL-6, IL-6R, IL-1RA, IL-1β, or GM-CSF antagonists, or a BTK inhibitor, within 7 days of randomization.
* Treatment with a JAK inhibitor within 30 days of randomization.
* Participants who are on long-term use of antirejection or immunomodulatory drugs.
* Pregnant or nursing (lactating) women.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2020-05-24 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (35):
  - Honor Health Research Institute, Scottsdale, Arizona
  - Sharp Memorial Hospital, San Diego, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Teradan Clinical Trials, Brandon, Florida
  - University of Florida, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Northshore University Health System, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Indiana University Health Central Indiana Cancer Centers, Indianapolis, Indiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Healthpartners Cancer Care Center - Regions Hospital, Saint Paul, Minnesota
  - Mercy Research, Springfield, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Njms Clinical Research Unit, Newark, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Kettering Cancer Care, Dayton, Ohio
  - Jefferson University Hospitals, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Allegheny Health Network, Wexford, Pennsylvania
  - St David'S Medical Center, Austin, Texas
  - University of Texas Health Science Center At Houston - McGovern Medical School, Houston, Texas
  - University of Texas Health Science Cente, San Antonio, Texas
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Aurora Research Institute, Milwaukee, Wisconsin
- Sbih City Hospital 15, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rein L, Calero K, Shah R, Ojielo C, Hudock KM, Lodhi S, Sadaka F, Bellam S, Palma C, Hager DN, Daniel J, Schaub R, O'Hayer K, Theodoropoulos NM. Randomized Phase 3 Trial of Ruxolitinib for COVID-19-Associated Acute Respiratory Distress Syndrome. Crit Care Med. 2022 Dec 1;50(12):1701-1713. doi: 10.1097/CCM.0000000000005682. Epub 2022 Oct 13. PMID 36226977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 33 study centers in the United States (29) and Russia (4), and 211 participants were enrolled and analyzed for efficacy.; 209 participants were analyzed for safety. Enrollment in this study was stopped early and was not due to safety reasons.
Pre-assignment Details: Participants were randomly assigned in a 2:2:1 ratio to receive ruxolitinib 5 mg BID, ruxolitinib 15 mg BID, or placebo for an initial treatment period of 14 days; participants randomly assigned to receive placebo were randomly assigned in a 1:1 ratio to receive placebo matching ruxolitinib 5 mg BID or placebo matching ruxolitinib 15 mg BID. Randomization was stratified by ARDS severity (severe vs mild/moderate at the time of randomization) and investigative site.
Groups:
- Ruxolitininb 15mg + Standard of Care: Ruxolitinib 15mg was administered BID approximately 12 hours apart without regard to food/feeding via enteric feeding tube or oral.
- Ruxolitinib 5mg + Standard of Care (SoC): Ruxolitinib 5mg was administered BID approximately 12 hours apart without regard to food/feeding via enteric feeding tube or oral.
- Placebo + Standard of Care (SoC): Matching Placebo was administered BID approximately 12 hours apart without regard to food/feeding via enteric feeding tube or oral.
Period: Overall Study
Arm/Group | Ruxolitininb 15mg + Standard of Care | Ruxolitinib 5mg + Standard of Care (SoC) | Placebo + Standard of Care (SoC)
Started | 77 | 87 | 47
Completed | 35 | 37 | 11
Not Completed | 42 | 50 | 36
Not completed — Death | 42 | 48 | 36
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized to the study.
Groups:
- Ruxolitininb 15mg + Standard of Care (SoC): Ruxolitinib 15mg was administered BID approximately 12 hours apart without regard to food/feeding via enteric feeding tube or oral.
- Total: Total of all reporting groups
Arm/Group | Ruxolitininb 15mg + Standard of Care (SoC) | Ruxolitinib 5mg + Standard of Care (SoC) | Placebo + Standard of Care (SoC) | Total
Number analyzed (Participants) | 77 | 87 | 47 | 211
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (12.92) | 63.6 (12.25) | 62.5 (13.34) | 63.4 (12.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 32 | 13 | 74
  Male | 48 | 55 | 34 | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 21 | 12 | 54
  Not Hispanic or Latino | 53 | 64 | 34 | 151
  Unknown or Not Reported | 3 | 2 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 3 | 3 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 12 | 5 | 26
  White | 57 | 61 | 31 | 149
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 11 | 8 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Have Died Due to Any Cause
Description: To evaluate the 28-day mortality rate of ruxolitinib 5 mg BID + SoC therapy and ruxolitinib 15 mg BID + SoC compared with placebo + SoC therapy, in participants with COVID-19-associated ARDS who require mechanical ventilation.
Time Frame: Study start to Day 29
Population: ITT population is defined according to the treatment assignment at the time of randomization regardless of the actual study drug the participant might take during his/her participation in the study.
Measure: Number; unit: Percentage
Arm/Group | Ruxolitininb 15mg + Standard of Care (SoC) | Ruxolitinib 5mg + Standard of Care (SoC) | Placebo + Standard of Care (SoC)
Number analyzed (Participants) | 77 | 85 | 47
Percentage | 50.6 | 52.9 | 70.2
Statistical Analysis 1: Comparison: Ruxolitininb 15mg + Standard of Care (SoC); Test type: Superiority; p = 0.0292, Mixed Models Analysis; logistic regression mixed model includes treatment group and ARDS severity as fixed covariates and investigational site as a random effect; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.201 to 1.028]
Statistical Analysis 2: Comparison: Ruxolitinib 5mg + Standard of Care (SoC); Test type: Superiority; p = 0.0280, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.171 to 1.023]

2. Secondary Outcome: Number of Ventilator Free Days
Description: Number of days participant did not require mechanical ventilation
Time Frame: Study start to Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ruxolitininb 15mg + Standard of Care (SoC) | Ruxolitinib 5mg + Standard of Care (SoC) | Placebo + Standard of Care (SoC)
Number analyzed (Participants) | 77 | 85 | 47
Days | 6.31 (9.047) | 4.92 (8.398) | 2.98 (7.228)

3. Secondary Outcome: Number of ICU Free Days
Description: Number of days participant is out of the ICU
Time Frame: Study start to Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ruxolitininb 15mg + Standard of Care (SoC) | Ruxolitinib 5mg + Standard of Care (SoC) | Placebo + Standard of Care (SoC)
Number analyzed (Participants) | 77 | 85 | 47
Days | 4.75 (7.716) | 4.00 (7.517) | 2.45 (6.362)

4. Secondary Outcome: Oxygen Free Days
Description: Number of days participant did not receive supplemental oxygen
Time Frame: Study start to Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ruxolitininb 15mg + Standard of Care (SoC) | Ruxolitinib 5mg + Standard of Care (SoC) | Placebo + Standard of Care (SoC)
Number analyzed (Participants) | 77 | 85 | 47
Days | 2.66 (6.073) | 2.98 (6.745) | 1.53 (4.690)

5. Secondary Outcome: Vasopressor Free Days
Description: Number of days without use of vasopressor therapy
Time Frame: Study start to Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ruxolitininb 15mg + Standard of Care (SoC) | Ruxolitinib 5mg + Standard of Care (SoC) | Placebo + Standard of Care (SoC)
Number analyzed (Participants) | 77 | 85 | 47
Days | 8.95 (11.738) | 7.53 (10.861) | 4.47 (9.322)

6. Secondary Outcome: Hospital Free Days
Description: Number of days Partcipant is out of the hospital
Time Frame: Study start to Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ruxolitininb 15mg + Standard of Care (SoC) | Ruxolitinib 5mg + Standard of Care (SoC) | Placebo + Standard of Care (SoC)
Number analyzed (Participants) | 77 | 85 | 47
Days | 2.09 (4.889) | 2.35 (5.259) | 1.38 (3.976)

7. Secondary Outcome: Percentage of Participants With at Least 2-point Improvement in the COVID-19 Ordinal Scale
Description: Participants with at least 2-point improvement at Day 15 and 29 based on participant state. The scale ranges from 0-8 with 0 being no clinical or virological evidence of infection and 8 being dead
Time Frame: Study start to Days 15 and 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ruxolitininb 15mg + Standard of Care (SoC) | Ruxolitinib 5mg + Standard of Care (SoC) | Placebo + Standard of Care (SoC)
Number analyzed (Participants) | 77 | 87 | 47
Percentage of Participants
  Day 15: number analyzed (Participants) | 77 | 85 | 47
  Day 15 | 22.1 [13.4 to 33.] | 15.3 [8.4 to 24.7] | 10.6 [3.5 to 23.1]
  Day 29: number analyzed (Participants) | 74 | 83 | 47
  Day 29 | 29.7 [19.7 to 41.5] | 25.3 [16.4 to 36.0] | 17.0 [7.6 to 30.8]

8. Secondary Outcome: Percentage of Participants With at Least 1-point Improvement in the COVID-19 Ordinal Scale
Description: Participants with at lest 1-point improvement in clinical status at Days 15 and 29 based on participant state. The scale ranges from 0-8 with 0 being no clinical or virological evidence of infection and 8 being dead
Time Frame: Study start to Days 15 and 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ruxolitininb 15mg + Standard of Care (SoC) | Ruxolitinib 5mg + Standard of Care (SoC) | Placebo + Standard of Care (SoC)
Number analyzed (Participants) | 77 | 87 | 47
Percentage of Participants
  Day 15: number analyzed (Participants) | 77 | 85 | 47
  Day 15 | 41.6 [30.4 to 53.4] | 32.9 [23.1 to 44.0] | 21.3 [10.7 to 35.7]
  Day 29 | 43.2 [31.8 to 55.3] | 32.5 [22.6 to 43.7] | 17.0 [7.6 to 30.8]

9. Secondary Outcome: Time to Improvement From Baseline Category to Earliest 1-point Improvement in the COVID-19 Ordinal Scale
Description: TIme to improvement compared to baseline. The scale ranges from 0-8 with 0 being no clinical or virological evidence of infection and 8 being dead
Time Frame: Study Start to Day 29
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Ruxolitininb 15mg + Standard of Care (SoC) | Ruxolitinib 5mg + Standard of Care (SoC) | Placebo + Standard of Care (SoC)
Number analyzed (Participants) | 50 | 49 | 20
Days | 0.91 [0.711 to 0.992] | 0.75 [0.614 to 0.867] | 0.61 [0.408 to 0.818]

10. Secondary Outcome: Percentage of Participants With the COVID-19 Ordinal Scale Reported
Description: Clinical status of participant at Day 29 based on participant state. The scale ranges from 0-8 with 0 being no clinical or virological evidence of infection and 8 being dead
Time Frame: Study start to Day 29
Population: ITT population is defined according to the treatment assignment at the time of randomization regardless of the actual study drug the participant might take during his/her participation in the study. Please note that in the 15mg BID arm, 3 participants were missing scale reporting on Day 29. In the 5mg BID, 2 participants were lost to follow-up, and 2 were missing scale reporting.
Measure: Number; unit: Percentage
Arm/Group | Ruxolitininb 15mg + Standard of Care (SoC) | Ruxolitinib 5mg + Standard of Care (SoC) | Placebo + Standard of Care (SoC)
Number analyzed (Participants) | 74 | 83 | 47
Percentage
  Score 0 = Uninfected | 0 | 4.6 | 0
  Score 1 = Ambulatory (no limitation of activities) | 2.6 | 0 | 2.1
  Score 2 = Ambulatory (limitation of activities) | 16.9 | 16.1 | 10.6
  Score 3 = Hospitalized/Mild Disease (no oxygen therapy) | 0 | 1.1 | 0
  Score 4 = Hospitalized/Mild Disease (oxygen therapy via mask or nasal prongs) | 9.1 | 1.1 | 4.3
  Score 5 = Hospitalized/Severe Disease (non-invasive ventilation or high-flow oxygen) | 3.9 | 4.6 | 0.0
  Score 6 = Hospitalized/Severe Disease (intubationand mechanical ventilization) | 10.4 | 8.0 | 2.1
  Score 7 = Hospitalized/Severe Disease (ventilation + additional organ support) | 2.6 | 8.0 | 10.6
  Score 8 - Death | 50.6 | 51.7 | 70.2

11. Secondary Outcome: Change in the COVID-19 9-point Ordinal Scale
Description: Change in the Clinical status of participant at Days 15 and 29 based on participant state. The scale ranges from 0-8 with 0 being no clinical or virological evidence of infection and 8 being dead
Time Frame: Study start to Days 15 and 29
Population: ITT population is defined according to the treatment assignment at the time of randomization regardless of the actual study drug the participant might take during his/her participation in the study. In the 15mg BID arm, 3 participants were missing scale reportingon Day 29. IN the 5mg BID, 2 participants were lost to follow-up, and 2 were missing scale reporting.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ruxolitininb 15mg + Standard of Care (SoC) | Ruxolitinib 5mg + Standard of Care (SoC) | Placebo + Standard of Care (SoC)
Number analyzed (Participants) | 77 | 87 | 47
Score on a Scale
  Change from Day 1 to Day 15: number analyzed (Participants) | 77 | 85 | 47
  Change from Day 1 to Day 15 | -0.4 (1.80) | -0.2 (1.73) | 0.6 (1.69)
  Change from Day 1 to Day 29: number analyzed (Participants) | 74 | 83 | 47
  Change from Day 1 to Day 29 | -0.5 (2.53) | -0.4 (2.57) | 0.4 (2.23)

12. Secondary Outcome: Change in SOFA Score
Description: Sequential Organ Failure Assessment (SOFA) score is a scoring system to determine the extent of a person's organ function or rate of failure. The score is based on 6 different scores, 1 each for the respiratory, cardiovascular, hepatic, coagulation, renal, and neurological systems. Each system gets a score from 0 (normal) to 4 (abnormal) and the sum of each score defines the final SOFA score, which 24 is the maximum score (high risk of morality) and 0 is the minimum score (low risk of mortality).
Time Frame: from baseline to Days 3, 5, 8, 11, 15, and 29
Population: ITT population is defined according to the treatment assignment at the time of randomization regardless of the actual study drug the participant might take during his/her participation in the study. Numbers of participants decreased after Day 1 because data was no longer collected if a patient was discharged from ICU and/or deceased.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Ruxolitininb 15mg + Standard of Care (SoC) | Ruxolitinib 5mg + Standard of Care (SoC) | Placebo + Standard of Care (SoC)
Number analyzed (Participants) | 77 | 87 | 47
Scores on a Scale
  Baseline - Day 1: number analyzed (Participants) | 74 | 87 | 46
  Baseline - Day 1 | 9.2 (2.35) | 9.6 (2.53) | 9.4 (2.69)
  Day 3: number analyzed (Participants) | 76 | 87 | 46
  Day 3 | -0.1 (2.77) | 0.4 (3.14) | 2.6 (5.89)
  Day 5: number analyzed (Participants) | 76 | 85 | 47
  Day 5 | 0.2 (4.27) | 0.7 (4.58) | 3.3 (6.60)
  Day 8: number analyzed (Participants) | 69 | 83 | 45
  Day 8 | 1.9 (6.77) | 2.0 (6.30) | 4.5 (7.87)
  Day 11: number analyzed (Participants) | 69 | 79 | 42
  Day 11 | 2.5 (7.64) | 2.0 (7.02) | 6.5 (8.26)
  Day 15: number analyzed (Participants) | 67 | 74 | 40
  Day 15 | 4.2 (9.24) | 4.1 (7.72) | 10.3 (7.89)
  Day 29: number analyzed (Participants) | 52 | 60 | 38
  Day 29 | 10.3 (8.54) | 10.4 (7.04) | 12.8 (5.41)

13. Secondary Outcome: Number and Percentage of Participants With Treatment-related Side Effects and Serious Adverse Events
Description: Treatment-emergent AEs are judged as related by the investigator or have a missing causality.
Time Frame: Study start to Day 29
Population: The safety population includes all participants who received at least 1 dose of ruxolitinib/placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitininb 15mg + Standard of Care (SoC) | Ruxolitinib 5mg + Standard of Care (SoC) | Placebo + Standard of Care (SoC)
Number analyzed (Participants) | 77 | 87 | 45
Participants
  Treatment-Emergent Adverse Events (TEAEs) | 22 | 23 | 11
  Serious TEAEs | 23 | 21 | 11

ADVERSE EVENTS:
Time Frame: Up to approximately 2 months.
Description: All-Cause Mortality was monitored in all randomized participants and Serious and Other Adverse Events were assessed only in participants who received the intervention (i.e. the safety population).
Groups:
- Ruxolitinib 15 mg BID: Ruxolitinib 15 mg BID
- Ruxolitinib 5 mg BID: Ruxolitinib 5 mg BID
- Placebo: Placebo
- Total: Total
Arm/Group | Ruxolitinib 15 mg BID | Ruxolitinib 5 mg BID | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 42/77 | 48/87 | 36/47 | 124/209
Serious Adverse Events (participants affected / at risk) | 23/77 | 21/87 | 11/45 | 55/209
Other Adverse Events (participants affected / at risk) | 35/77 | 46/87 | 21/45 | 102/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib 15 mg BID (N=77) | Ruxolitinib 5 mg BID (N=87) | Placebo (N=45) | Total (N=209)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 3 (4) | 1 (1) | 5 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 5 (5)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 2 (3) | 4 (4) | 2 (2) | 8 (9)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 4 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Strongyloidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Torsade de pointes (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vascular device infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib 15 mg BID (N=77) | Ruxolitinib 5 mg BID (N=87) | Placebo (N=45) | Total (N=209)
Alanine aminotransferase increased (Investigations) | 9 (9) | 12 (13) | 5 (5) | 26 (27)
Anaemia (Blood and lymphatic system disorders) | 12 (13) | 21 (23) | 9 (9) | 42 (45)
Anxiety (Psychiatric disorders) | 6 (6) | 4 (4) | 1 (1) | 11 (11)
Aspartate aminotransferase increased (Investigations) | 10 (10) | 11 (12) | 3 (3) | 24 (25)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 5 (6) | 3 (3) | 9 (10)
Bacteraemia (Infections and infestations) | 1 (1) | 5 (5) | 0 (0) | 6 (6)
Constipation (Gastrointestinal disorders) | 5 (5) | 4 (4) | 2 (2) | 11 (11)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (5) | 3 (4) | 10 (13)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 8 (9) | 1 (1) | 12 (14)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 3 (3) | 10 (10)
Hypermagnesaemia (Metabolism and nutrition disorders) | 5 (7) | 4 (4) | 1 (1) | 10 (12)
Hypernatraemia (Metabolism and nutrition disorders) | 8 (13) | 7 (8) | 7 (7) | 22 (28)
Hypertension (Vascular disorders) | 5 (5) | 11 (12) | 5 (5) | 21 (22)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 7 (7) | 4 (4) | 12 (12)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (11) | 9 (11) | 4 (4) | 22 (26)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 3 (4) | 8 (10)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5) | 6 (8) | 2 (2) | 13 (15)
Hypotension (Vascular disorders) | 4 (5) | 3 (3) | 2 (2) | 9 (10)
Lymphocyte count decreased (Investigations) | 3 (5) | 4 (7) | 3 (4) | 10 (16)
Oedema peripheral (General disorders) | 2 (2) | 5 (6) | 0 (0) | 7 (8)
Pneumonia staphylococcal (Infections and infestations) | 5 (5) | 2 (2) | 1 (1) | 8 (8)
Pyrexia (General disorders) | 2 (2) | 5 (7) | 4 (4) | 11 (13)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (4) | 5 (6) | 3 (3) | 11 (13)
Vomiting (Gastrointestinal disorders) | 5 (10) | 4 (5) | 1 (1) | 10 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT04377620/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT04377620/SAP_001.pdf